CLINICAL TRIAL: NCT04151849
Title: Complementary Effects of New Diabetes Medications on Adrenal Function and Intestinal Microbiota
Brief Title: Effects of Diabetes Medications on Adrenal Function and Intestinal Microbiota
Status: Completed | Type: Observational
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Vallo Volke, Professor, University of Tartu
Other Study IDs: 290/T-20
Record Dates: First submitted 2019-10-29; First posted 2019-11-05 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes
Keywords: GLP-1 receptor agonist; SGLT-2 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- GLP-1 receptor agonist treatment: Patients starting treatment with any molecule belonging to the class of GLP-1 receptor agonist.
  Interventions: Drug: GLP-1 receptor agonist
- SGLT-2 inhibitor treatment: Patients starting treatment with any molecule belonging to the class of SGLT-2 inhibitors.
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: GLP-1 receptor agonist — Treatment with GLP-1 agonist for up to 1 year.
  Groups: GLP-1 receptor agonist treatment
Drug: SGLT2 inhibitor — Treatment with SGLT2 inhibitor for up to 1 year
  Groups: SGLT-2 inhibitor treatment

SUMMARY:
The primary aim of this observational study is to describe the effects of glucagon-like peptide-1 (GLP-1) receptor agonists and Sodium-Glucose Co-transporter 2 inhibitors ( SGLT-2 inhibitors) on adrenal function. Secondary endpoint is change in intestinal microbiota.

DETAILED DESCRIPTION:
This is an observational study conducted in patients with type 2 diabetes starting treatment with either GLP-1 receptor agonist or sodium-glucose cotransporter-2 (SGLT-2) inhibitor.

Planned study cohort consists of 60 patients: 30 patients starting GLP-1 receptor agonist treatment and 30 patients starting SGLT-2 inhibitor treatment. All patients must have metformin as background therapy. All other diabetes medications are allowed.

Patients are tested before starting treatment, at 1 month (stool sample only), 3 months and 12 months after starting treatment. The primary endpoint is change in overnight urinary aldosterone corrected for creatinine.

Secondary endpoint is change in intestinal microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Type 2 diabetes
* HbA1c < 10%
* BMI >32
* Daily dose of metformin 1,5 g or more.
* No change in diabetes treatment at least 90 days before starting the study.
* Never used SGLT-2 inhibitors or/and GLP-1 receptor agonist.
* Tested negative to glutamic acid decarboxylase 65 autoantibodies.

Exclusion Criteria:

* Pregnancy and lactation.
* Use of systemic antibiotic treatment < 60 days before starting the study.
* Use of spironolactone < 60 days before starting the study.
* Use of oral contraceptives or hormonal replacement therapy.
* Use of immunosuppressive drug
* Heart failure New York Heart Association III-IV
* Severe liver disease.
* Malignant disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes who need treatment intensification with SGLT-2 inhibitor or GLP-1 receptor agonist.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Urinary aldosterone at 3 months | 3 months
  Overnight urinary aldosterone compared to pretreatment level.

SECONDARY OUTCOMES:
Change in gastrointestinal microbiota. | At 1 month after starting treatment, at 3 months and 12 months.
  Fecal microbiota will be compared to pre-treatment sample.
Urinary aldosterone at 12 months | 12 months
  Overnight urinary aldosterone at 12 months compared to pretreatment level.

OTHER OUTCOMES:
Serum adrenocorticotropic hormone | At 3 months and 12 months.
  Change in adrenocorticotropic hormone in serum compared to pretreatment level.
Plasma cortisol | At 3 months and 12 months.
  Change in plasma cortisol compared to pretreatment level
Urinary cortisol | At 3 months and 12 months.
  Change in overnight urinary cortisol compared to pretreatment level.
Plasma aldosterone | At 3 months and 12 months.
  Change in plasma aldosterone compared to pretreatment level.
Plasma renin | At 3 months and 12 months.
  Change in plasma renin compared to pretreatment level.
Serum sodium | At 3 months and 12 months.
  Change in serum sodium compared to pretreatment level.
Serum potassium | At 3 months and 12 months.
  Change in serum potassium compared to pretreatment level.
Glycated hemoglobin A1c | At 3 months and 12 months.
  Change in glycated hemoglobin A1c compared to pretreatment level.
Ceruloplasmin | At 3 months and 12 months.
  Change in plasma ceruloplasmin compared to pretreatment level.
Ferritin | At 3 months and 12 months.
  Change in plasma ferritin compared to pretreatment level.

CONTACTS AND LOCATIONS:
Overall Officials: Vallo Volke, MD, PhD, Principal Investigator — University of Tartu, Institute of Biomedicine and Translational Medicine
Locations (1):
- Tartu University Hospital, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No